CLINICAL TRIAL: NCT05173883
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of a Single Subcutaneous Injection of CU-20401 in Chinese Healthy Population
Brief Title: A Phase 1 Clinical Study of CU-20401 in Chinese Healthy Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cutia Therapeutics（Wuxi）Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CU-20401-102
Record Dates: First submitted 2021-11-30; First posted 2021-12-30 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Healthy Subjects
Keywords: safty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- A cohort of CU-20401 (Experimental): Subcutaneous injection in the subcutaneous fat area，0.2ml of CU-20401, 6 injections，0.04mg/ml（A1)，0.075mg/ml(A2)，0.15mg/ml(A3)
  Interventions: Drug: injection ，CU-20401
- B cohort of CU-20401 (Experimental): Subcutaneous injection in the subcutaneous fat area，0.2ml of CU-20401, 12 injections，0.075mg/ml（B1)，0.10mg/ml(B2)
  Interventions: Drug: injection ，CU-20401
- C cohort and D cohort of CU-20401 (Experimental): Subcutaneous injection in the subcutaneous fat area，0.2ml of CU-20401, 24 injections，0.075mg/ml（C1)，0.10mg/ml(C2)，0.12mg/ml(D2),
  Interventions: Drug: injection ，CU-20401
- A cohort of placebo (Placebo Comparator): Subcutaneous injection in the subcutaneous fat area，0.2ml of placebo, 1 injections，0.04mg/ml（A1)，0.075mg/ml(A2)，0.15mg/ml(A3)
  Interventions: Drug: injection ，placebo
- B cohort of placebo (Placebo Comparator): Subcutaneous injection in the subcutaneous fat area，0.2ml of placebo, 1 injections，0.075mg/ml（B1)，0.10mg/ml(B2)
  Interventions: Drug: injection ，placebo

INTERVENTIONS:
Drug: injection ，CU-20401 — Subcutaneous injection，cohort A 6 sites
  Other Names: test group administration
  Arms: A cohort of CU-20401; B cohort of CU-20401; C cohort and D cohort of CU-20401
Drug: injection ，placebo — Subcutaneous injection，just one site
  Other Names: Control group administration
  Arms: A cohort of placebo; B cohort of placebo

SUMMARY:
This is an open-label, Part I/2/3/4 Phase 1 clinical study to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of a single subcutaneous injection of CU-20401 in healthy Chinese population, and to recommend an appropriate dose for subsequent clinical studies.

DETAILED DESCRIPTION:
In Part 1, 3 dose groups (dose group A1) were prespecified : 0.04 mg/dose; Dose Group A2 : 0.075 mg/dose; Dose Group A3 : 0.15 mg/dose). Eligible subjects were enrolled in the order from the low dose group to the high dose group (A1 → A2 → A3), and all subjects in the first dose group completed dosing.All examinations (vital signs, physical examination, laboratory tests, 12-lead ECG, abdominal wall color ultrasonography, etc.) will be performed during the dosing observation period and the follow-up period. Only after the investigator confirms that no subject meets the criteria for discontinuation of escalation, the next dose group can be started. Two subjects will be enrolled in each dose group for at least 24 h, and the remaining 4 subjects will not be enrolled until no safety events have occurred.

Eligible subjects were sequentially enrolled in Dose Group B1 (0.075 mg/dose) and Dose Group B2 (0.10 mg/dose) to receive the established dose. All examinations (vital signs, physical examination, laboratory tests, 12-lead ECG, abdominal B-ultrasound, etc.) will be performed during the dosing observation period .All subjects may enter Part 3 of the study after the investigator confirms that all subjects have completed the visit on D7 and no intolerable safety events have occurred. The subject continued to receive subsequent follow-up (D14/D21/D29).

Eligible subjects were sequentially enrolled in dose group C1 (0.075 mg/dose) and dose group C2 (0.10 mg/dose) to receive the established dose; doses were administered bilaterally with 12 injections on each side. All examinations (vital signs, physical examination, laboratory tests, 12-lead ECG, abdominal B-ultrasound, etc.) were performed during the dosing observation period. During the follow-up period, a visit on D7/D14/D21/D29/D56/D84 was required. After subjects in Part III have completed at least the visit on D29, and no intolerable safety events have occurred, Part IV of the study may be conducted in consultation with the investigator and the sponsor.

Based on the available data, a dose of 0.12 mg/dose is tentatively proposed for Part 4 of the study, administered bilaterally with 12 injections on each side. The study procedures are the same as Part III.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 to 50 years (including boundary values);
2. Abdominal skinfold thickness ≥ 4 cm;
3. Inquiries such as medical history, physical examination, vital signs, 12-lead electrocardiogram, chest X-ray, B-ultrasound and laboratory tests are normal or abnormal, and are not clinically significant as judged by the investigator;
4. Female subjects had a negative blood pregnancy test; The subject has no sperm or egg donation plan within 90 days after signing the informed consent form; Subjects have no fertility plan and voluntarily take effective contraceptive measures during the study and within 90 days after dosing:

   1. True abstinence;
   2. Use of double barrier contraception, i.e. use of spermicide or cervical cap or vaginal diaphragm while using condom;
   3. Intrauterine device;
   4. Tubal ligation or hysterectomy;
   5. Partner sterilization for male or female subjects.
5. Fully understand the purpose, requirements and risks of this study, voluntarily participate in the clinical trial and sign a written informed consent form, and can complete the entire study process in accordance with the requirements of the trial.

   -

Exclusion Criteria:

1. Patients with the following diseases suggested by screening examination:

   including but not limited to respiratory system, circulatory system, digestive system, blood system, endocrine system, immune system, skin system, psychoneurological system, otology and other related diseases; subjects who, as judged by the investigator, may increase relevant risks, or may affect the study results, and are not suitable for participation in this study
2. Allergic constitution, history of allergy to collagenase or components of the study drug or its excipients;
3. Received collagenase treatment within 6 months prior to screening;
4. Received surgery, instrumental lipolysis, laser therapy within 12 months prior to screening, or planned surgery, lipolysis, laser therapy, etc., during the study;
5. Having undergone liposuction surgery or taking any medication or health care product for the purpose of weight loss within six months prior to screening;
6. Participated in clinical trials of other study drugs within 3 months prior to screening;
7. Hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, treponema pallidum antibody (Anti-TP) test positive;
8. Donation of blood within 3 months prior to screening includes component blood or massive blood loss (≥ 400 mL); those who receive blood transfusion or use blood products;
9. For patients with bleeding abnormalities or currently receiving antiplatelet therapy (except for patients taking aspirin ≤ 150 mg per day) or anticoagulant therapy;
10. Significant changes in abnormal diet or eating habits within 30 days prior to screening;
11. Tattoos or scars, skin lesions (such as abrasions, etc.), skin infections (such as dermatitis, etc.) at the intended operation site affect the drug administration or the observer;
12. History of drug abuse within 6 months prior to screening, or positive urine drug abuse screening;
13. Smoking more than 5 cigarettes per day within 3 months prior to screening, or unable to stop using any tobacco products during the trial;
14. Alcoholics or regular drinkers within 3 months prior to the trial, i.e., more than 21 units of alcohol per week (1 unit = 360mL of beer or 45 mL of spirits with 40% alcohol or 150 mL of wine), or those with a positive alcohol breath test;
15. Current or former drug user;
16. Vaccinated within 1 month prior to screening;
17. Suffering from other acute or chronic medical or psychiatric disorders that, as judged by the investigator, are not suitable for participation in this study, may increase the risks associated with participation in this study, or may interfere with the interpretation of the study results;
18. Lactating and pregnant women;
19. Subjects unable to undergo MRI;
20. Other conditions judged by the investigator to be inappropriate for participation in this study.

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Abdominal fat volume | Day 29/56/84
  The proportion of subjects with at least a 10% reduction from baseline in abdominal (dosing area) fat volume was evaluated using MRI; (Part II is limited to D29 and Part III and IV are on D29/56/84)

SECONDARY OUTCOMES:
Abdominal fat thickness | Day 29
  The thickness of abdominal fat on day 29 changes from baselinefat thickness in the abdominal B-ultrasound administration area in all subjects receiving the investigational product, and the relationship between the administered dose and efficacy will be assessed.

OTHER OUTCOMES:
the proportion of changes from baseline and changes in abdominal (dosing area) fat volume. | Day 29/56/84
  MRI was used to evaluate the proportion of changes from baseline and changes in abdominal (dosing area) fat volume. (Part II is limited to D29 and Part III and IV are on D29/56/84)

CONTACTS AND LOCATIONS:
Overall Officials: TANIA LI, MM, Study Director — CUTIA
Locations (1):
- Shanghai Xuhui Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No